CLINICAL TRIAL: NCT01688167
Title: Increasing Availability and Acceptability of Circumcision in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen Weiss, Research Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20110290; R01MH095539 (NIH)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: HIV
Keywords: HIV; Male circumcision; Sexual risk reduction; Stages of change

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): Experimental condition clinics offer the MC and sexual risk reduction intervention: four group counseling sessions focused on male circumcision and sexual risk reduction.
  Interventions: Behavioral: MC and sexual risk reduction
- Standard of Care (No Intervention): Male participants in the standard of care control condition CHCs will receive counseling per the VCT protocol guidelines. Participants will attend four video-based time-equivalent "attention-control" group sessions on endemic disease prevention strategies (e.g., TB, malaria, cholera, waterborne diseases). Female partners will be invited to participate in a similar four session program devoted to endemic disease risk reduction.
- Observational (No Intervention): 3 CHC sites will be randomly assigned as "observation only;" only aggregated clinic VCT and circumcision data will be collected.

INTERVENTIONS:
Behavioral: MC and sexual risk reduction — Four group counselling sessions focused on male circumcision and sexual risk reduction
  Arms: Intervention

SUMMARY:
This study proposes to balance supply and demand of male circumcision through a systematic scale-up of coordinated biomedical surgical and behavioral counseling services. The study will compare the combined biobehavioral sexual risk reduction intervention to the standard of care, which focuses exclusively on the provision of circumcision services alone, with the goal of optimizing both local and national HIV prevention efforts.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative
* Uncircumcised male
* 18+ years of age
* Able to understand and sign informed consent in English, Bemba, or Nyanja
* Have not requested male circumcision services at the time of or following VCT
* Female partners of enrolled males are invited to participate

Exclusion Criteria:

* Men seeking circumcision services are not eligible for this study
* Men with genital abnormalities requiring MC, e.g. balanitis (inflammation of the preputial skin), posthitis (inflammation of the glans penis; common in patients with diabetes), phimosis (scarring of the distal margins of the foreskin) resulting from chronic balanitis, paraphimosis (the inability to pull the retracted foreskin back over the glans) or diseases of the foreskin, including localized carcinoma are not eligible for this study
* Men with congenital or acquired penile abnormalities that require the preputial skin for generative repair, such as hypospadias (urethra exits from underside of penis) are not eligible to participate
* Participants unable to provide informed consent will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1468 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in likelihood of undergoing male circumcision across the study using stages of change model | Baseline, Average of 1 month post-baseline, 6 month and 12 month follow-up
  Readiness to undergo male circumcision will be assessed using the stages of change model (pre-contemplation, contemplation, preparation, action, maintenance). Intervention and attention control conditions will be compared at baseline, immediately following intervention, and 6 and 12 months post-intervention.

SECONDARY OUTCOMES:
Uptake of male circumcision | From the date of study enrollment to the date male circumcision is performed or study completion.
  To determine if participants in the sexual risk reduction/MC promotion intervention (experimental condition) will be more likely to shift to the "Action" stage (undergo circumcision), in comparison with participants having identical MC services available plus usual care (attention control condition).

OTHER OUTCOMES:
Male and female condom use post male circumcision | 3 months after undergoing male circumcision
  To determine whether MC will significantly affect the maintenance of safer sexual practices ("risk compensation") in the experimental group as compared to the attention control group

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Weiss, PhD, Study Chair — University of Miami
Locations (1):
- University of Zambia Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Background] Weiss SM, Zulu R, Jones DL, Redding CA, Cook R, Chitalu N. The Spear and Shield intervention to increase the availability and acceptability of voluntary medical male circumcision in Zambia: a cluster randomised controlled trial. Lancet HIV. 2015 May;2(5):e181-9. doi: 10.1016/S2352-3018(15)00042-9. PMID 26120594
- [Background] Jones DL, Lopez M, Simons H, Diaz-Gloster M, Tobin JN, Weiss SM. Translation of a comprehensive health behavior intervention for women living with HIV: the SMART/EST Women's Program. Transl Behav Med. 2013 Dec;3(4):416-25. doi: 10.1007/s13142-013-0213-4. PMID 24294330
- [Background] Jones D, Weiss S, Chitalu N. HIV Prevention in Resource Limited Settings: A Case Study of Challenges and Opportunities for Implementation. Int J Behav Med. 2015 Jun;22(3):384-92. doi: 10.1007/s12529-014-9397-3. PMID 24604206
- [Background] Cook R, Jones D, Redding CA, Zulu R, Chitalu N, Weiss SM. Female Partner Acceptance as a Predictor of Men's Readiness to Undergo Voluntary Medical Male Circumcision in Zambia: The Spear and Shield Project. AIDS Behav. 2016 Nov;20(11):2503-2513. doi: 10.1007/s10461-015-1079-x. PMID 25931242
- [Background] Redding CA, Jones D, Zulu R, Chitalu N, Cook R, Weiss SM. Stages of Change for Voluntary Medical Male Circumcision and Sexual Risk Behavior in Uncircumcised Zambian Men: The Spear and Shield Project. Int J Behav Med. 2015 Dec;22(6):799-806. doi: 10.1007/s12529-015-9485-z. PMID 25896876